CLINICAL TRIAL: NCT03104361
Title: Intravesical Injections of Platelet-Rich Plasma (PRP) in Treatment of Interstitial Cystitis Refractory to Conventional Treatment - A Prospective, Clinical Trial
Brief Title: Platelet-Rich Plasma (PRP) Injection in Treatment of Interstitial Cystitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chairman, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCGH10548A
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Interstitial Cystitis
Keywords: intersitial cystitis; Bladder pain syndrome; Intravesical treatment
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Intravesicai injection of platelet-rich plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet-rich plasma treatment arm (Experimental): Patients who meet all eligible requirements for entry into the study will be treated with intravesical injection of PRP (extracted from 50ml whole blood ) at 20 sites
  Interventions: Biological: Platelet-Rich Plasma

INTERVENTIONS:
Biological: Platelet-Rich Plasma — Patients who meet all eligible requirements for entry into the study will be treated with intravesical injection of PRP (extracted from 50ml whole blood ) at 20 sites
  Other Names: PRP

SUMMARY:
Interstitial cystitis/painful bladder syndrome (IC/PBS) is a debilitating chronic disease of unknown etiology characterized by urgency frequency and suprapubic pain at full bladder. Current treatments are usually unsuccessful in completely eradicating bladder pain and increasing bladder capacity. Autologous platelet-rich plasma (PRP) is growing in popularity as a therapy to augment wound healing, speed the recovery from muscle and joint injuries, and enhance recovery after surgical repair. PRP is extremely rich in growth factors and cytokines, which regulate tissue reconstruction and has been studied extensively among trauma patients and trauma experimental models. Tissue regeneration can be improved by local application of autologous bone marrow derived progenitor cells and PRP. This clinical trial attempts to use autologous PRP in treatment of interstitial cystitis refractory to currently available medical treatment or intravesical therapy. The results of this study might provide clinical evidence for a novel therapeutic regimen in the treatment of IC/PBS.

DETAILED DESCRIPTION:
Background: Interstitial cystitis/painful bladder syndrome (IC/PBS) is a debilitating chronic disease of unknown etiology characterized by urgency frequency and suprapubic pain at full bladder. Current treatments are usually unsuccessful in completely eradicating bladder pain and increasing bladder capacity. Autologous platelet-rich plasma (PRP) is growing in popularity as a therapy to augment wound healing, speed the recovery from muscle and joint injuries, and enhance recovery after surgical repair. PRP is extremely rich in growth factors and cytokines, which regulate tissue reconstruction and has been studied extensively among trauma patients and trauma experimental models. Tissue regeneration can be improved by local application of autologous bone marrow derived progenitor cells and PRP.

Aim: This clinical trial attempts to use autologous PRP in treatment of interstitial cystitis refractory to currently available medical treatment or intravesical therapy. The results of this study might provide clinical evidence for a novel therapeutic regimen in the treatment of IC/PBS.

Setting: Department of Urology, Buddhist Tzu Chi General Hospital.

Materials and Methods: A total of 30 patients with IC/PBS who have failed conventional treatments for at least 6 months will be enrolled in this study. A diagnosis of IC/PBS has been established based on characteristic symptoms and cystoscopic findings of glomerulations, petechia, or mucosal fissures after hydrodistention. All patients have been treated with at least two types of treatment modalities including oral PPS, intravesical instillation of heparin, hyaluronic acid, or tricyclic antidepressant for at least 6 months but the symptoms remained unchanged or relapsed. All patients should have IC symptoms for at least 6 months, and proven to have grade 1 diffused glomerulations after cystoscopic hydrodistention (HD) within recent 1 year without Hunner's lesion. Eligible patients will be admitted for the treatment. The patients will receive intravesical injection of 12ml PRP (extracted from 50ml of patient's own whole blood) followed by cystoscopic hydrodistention under intravenous general anesthesia in the operation room. The procedure will repeat every one month for a total of four treatments. Blood (10ml) and urine samples (30ml) will be collected before intravesical PRP injection and at 4, 12 and 24 weeks after PRP injection.

Assessment: Primary end-point is the change of the O'Leary-Sant symptom score (including ICSI and ICPI) from baseline to 6 months after the first treatment day. Secondary endpoints include VAS, daily frequency, nocturia and FBC as record in 3-day voiding diary, Qmax, vided volume, PVR and global response assessment (GRA). Four visits are required at baseline screening (before first treatment) (V1), 1 month after the first treatment (V2, primary end-point), 4 weeks after the fourth treatment (V3), 24 weeks after the first treatment (V4, secondary end-point).

Urine samples will be collected at each time-point for NGF and cytokines tests. Bladder biopsy will be performed at baseline and 6 months after the first treatment day if possible.

Adverse events including UTI, AUR, large PVR (>150ml), dysuria and micturition pain will be recorded

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age of 20 years old or above
2. Patients with symptoms of frequency, urgency, nocturia, and/or bladder pain.
3. Proven to have glomerulations (at least grade 2) by cystoscopic hydrodistention under anesthesia in recent 1 year
4. Free of active urinary tract infection
5. Free of bladder outlet obstruction on enrolment
6. Free of overt neurogenic bladder dysfunction and limitation of ambulation
7. Patient or his/her legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

1. Hunner's lesion proven by cystoscopy
2. Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
3. Patients with bladder outlet obstruction on enrollment
4. Patients with postvoid residual >250ml
5. Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
6. Patients have laboratory abnormalities at screening including: ALT> 3 x upper limit of normal range, AST> 3 x upper limit of normal range; Patients have abnormal serum creatinine level > 2 x upper limit of normal range
7. Patients with any contraindication to be urethral catheterization during treatment
8. Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
9. Patients with any other serious disease considered by the investigator not in the condition to enter the trial
10. Patient had received intravesical onabotulinumtoxinA treatment for IC within recent 3 months
11. Patients participated investigational drug trial within 1 month before entering this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
O'Leary-Sant Symptom Score | from baseline to 1 month after the first treatment day
  1. Change of the O'Leary-Sant symptom score (including IC symptom index, ICSI, and IC problem index, ICPI)

SECONDARY OUTCOMES:
Visual analog score (VAS) for pain | from baseline to 6 months after the treatment day
  Net change of the Visual analog score (VAS) for pain (from 0 to 10)
Functional bladder capacity (FBC) | from baseline to 6 months after the treatment day
  Net change of functional bladder capacity
Voiding frequency | from baseline to 6 months after the treatment day
  Net change of voiding frequency at daytime and voiding frequency at night time as record in 3-day voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng kuo, M.D, Principal Investigator — Department of Urology, Buddhist TzuChi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers

REFERENCES:
- [Derived] Jiang YH, Kuo YC, Jhang JF, Lee CL, Hsu YH, Ho HC, Kuo HC. Repeated intravesical injections of platelet-rich plasma improve symptoms and alter urinary functional proteins in patients with refractory interstitial cystitis. Sci Rep. 2020 Sep 16;10(1):15218. doi: 10.1038/s41598-020-72292-0. PMID 32939046